CLINICAL TRIAL: NCT04141475
Title: Evaluation of Alpha-Lipoic Acid in Diabetic Cardiomyopathy
Acronym: CARDIALA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no patient recruitment
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-PP-07
Record Dates: First submitted 2019-10-25; First posted 2019-10-28 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Diabetic Cardiomyopathies
MeSH Terms: conditions — Diabetic Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alpha-Lipoic Acid group (Active Comparator)
  Interventions: Dietary Supplement: Physiomance acide lipoïque gold
- placebo group (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo - Physiomance acide lipoïque gold

INTERVENTIONS:
Dietary Supplement: Physiomance acide lipoïque gold — 1 capsule of 300 mg in the morning outside a meal and 1 capsule of 300 mg in the evening outside a meal during 12 weeks
  Arms: Alpha-Lipoic Acid group
Dietary Supplement: Placebo - Physiomance acide lipoïque gold — 1 capsule of 300 mg in the morning outside a meal and 1 capsule of 300 mg in the evening outside a meal during 12 weeks
  Arms: placebo group

SUMMARY:
The heart has the ability to respond to different patho-physiological conditions by adapting its energy metabolism. In diabetic subjects, the myocardium uses only fatty acids as a substrate. This is the cause of diabetic cardiomyopathy (DCM). The activation of the transcription factor PPARβ/δ allows a good use of fatty acids. The staff have demonstrated that alpha lipoic acid (AαL), a molecule with antioxidant properties present in food supplements and in certain foods (broccoli, cabbage, offal...), induces the expression of PPARβ/δ in skeletal muscle and thus increases the activity of this transcription factor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult age ≥ 18 years
* patient with diagnosed type 2 diabetes (history of pathological hyperglycemia according to WHO and HbA1c standards >7% or ongoing treatment with oral antidiabetic agents).
* Patients with stable cardiomyopathy (no hospitalization in cardiology in the month before inclusion) with a left ventricular ejection fraction (LVEF) <50%.
* patient who has signed an informed consent form
* For women of childbearing age: effective contraception followed for at least 3 months before the start of the study and agreeing to keep it for the duration of the study.
* affiliation to a social security scheme.

Exclusion Criteria:

subjects:

* With a coronary event in the year before inclusion.
* With symptoms of cardiac ischemia at inclusion.
* Pregnant or breastfeeding woman
* Severe renal insufficiency
* Using antioxidant molecules in the 6 months prior to inclusion.
* Using drugs that can activate PPARs (Fibrates, Telmisartan, Enalaprilat).
* Using anti-inflammatory drugs.
* Suffering from acute infectious diseases and inflammatory diseases.
* Hypersensitivity or a history of hypersensitivity reaction to gadoteric acid, meglumine or any drug containing gadolinium.

Non-inclusion criteria related to MRI:

* with an implanted vascular stent less than 6 weeks before the examination;
* carrier of an implanted biomedical device deemed "not safe" or "unsafe" in the list: http://www.mrisafety.com/TheList_search.asp;
* Beneficiary of an acquisition procedure that does not respect the conditions required by "conditional" use in a subject carrying an implanted biomedical material considered "conditional" in the list: http://www.mrisafety.com/TheList_search.asp;
* carrier of a ferromagnetic intraocular or intracranial foreign body close to the nerve structures;
* carrying biomedical equipment such as a cardiac, neural or sensory pacemaker (cochlear implant) or a ventricular bypass valve without medical and paramedical supervision trained to perform MRI in these subjects;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
change of LVEF between before and after 12 weeks of treatment | 12 weeks
  percentage of blood ejection before and after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Nice Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No